CLINICAL TRIAL: NCT00232440
Title: A Study to Examine the Reproducibility of an Immobilization Device (BodyFIX ) to Deliver High Precision Radiation Therapy for Patients With Hodgkin's Disease or Non-Hodgkin's Lymphoma
Brief Title: Reproducibility of an Immobilization Device (BodyFIX) - Hodgkins/Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHN REB 02-0526-C
Record Dates: First submitted 2005-10-03; First posted 2005-10-04 (Estimated); Last update posted 2010-08-11 (Estimated); Status verified 2010-08

CONDITIONS: Hodgkin's Disease; Lymphoma, Non-Hodgkin
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin

INTERVENTIONS:
Device: BodyFIX

SUMMARY:
Radiation therapy has a well-established role in the treatment of Hodgkin's Disease and non-Hodgkin's Lymphoma. With technological developments, 3-D Dimensional (3D) planning has evolved as a highly precise treatment planning option. High-precision radiation therapy has the potential for more accurate dose delivery to the tumour volume and can result in a greater sparing of normal tissue. An important component of safe radiotherapy delivery is the feasibility and reproducibility of current and new immobilization devices for highly conformal treatment.

The purpose of this study is to determine the reproducibility of an immobilization device known as BodyFIX(TM) using conventional treatment techniques.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing curative or palliative treatment in whom it is considered that immobilization of part or all of an anatomical region would be of benefit to their care.

Exclusion Criteria:

* Any case where ideal treatment may be compromised with use of immobilization method.
* If the patient has any social issues, language barriers resulting in difficulties comprehending the nature of the study, or poor performance status, that could compromise compliance with the study guidelines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2003-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
The primary outcome for the study is the average deviation in set-up.

CONTACTS AND LOCATIONS:
Overall Officials: Alex Sun, MD, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- University Health Network, Toronto, Ontario, Canada